CLINICAL TRIAL: NCT01464879
Title: A Phase 2, Open-Label, Sequential Dose Escalation Study in Adult Hypogonadal Males to Evaluate the Pharmacokinetics of Three Volumes of FE 999303 (Testosterone Gel), Applied to the Shoulder/Upper Arm, Using an Applicator Compared With Hand Application
Brief Title: A Clinical Study to Evaluate the Pharmacokinetics of Testosterone Gel Using an Applicator
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000024
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Hypogonadal Males

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Testosterone 2.50 mL (hand) (Experimental): Subjects in this arm self-applied two strokes (2.50 mL) of testosterone gel by hand, one stroke to the shoulder/upper arm and a second stroke to the contralateral shoulder/upper arm every day for seven days.
  Interventions: Drug: Testosterone Gel (FE 999303)
- Testosterone 1.25 mL (applicator) (Experimental): Subjects in this arm self-applied one stroke (1.25 mL) of testosterone gel by applicator to the shoulder/upper arm every day for seven days.
  Interventions: Drug: Testosterone Gel (FE 999303)
- Testosterone 2.50 mL (applicator) (Experimental): Subjects in this arm self-applied two strokes (2.50 mL) of testosterone gel by applicator, one stroke to the shoulder/upper arm and a second stroke to the contralateral shoulder/upper arm every day for seven days.
  Interventions: Drug: Testosterone Gel (FE 999303)
- Testosterone 3.75 mL (applicator) (Experimental): Subjects in this arm self-applied three strokes (3.75 mL) of testosterone gel by applicator, one stroke to the shoulder/upper arm and a second stroke to the contralateral shoulder/upper arm and a third stroke to the first shoulder/upper arm, every day for seven days.
  Interventions: Drug: Testosterone Gel (FE 999303)

INTERVENTIONS:
Drug: Testosterone Gel (FE 999303)

SUMMARY:
This is a Phase 2 clinical trial in adult hypogonadal males with baseline morning serum testosterone concentrations <300 ng/dL. The purpose of this study is to evaluate the pharmacokinetics of FE 999303, delivered using an applicator in comparison to hand application

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75
* History of hypogonadism
* In good health based on medical history, physical examination, and clinical laboratory tests
* Serum testosterone deficiency
* One or more symptom(s) of testosterone deficiency (i.e. fatigue, reduced libido, or reduced sexual functioning)
* Body mass index (BMI) between 18 and 35 kg/m^2
* All screening lab tests within 20% of the normal range (exceptions are liver function tests)
* HIV, Hepatitis B and C negative

Exclusion Criteria:

* Previous use of FE 999303
* Prostate cancer
* Breast carcinoma, patient or partner
* Palpable prostatic mass(es)
* Serum PSA levels ≥3 ng/dL
* Chronic use of any drug of abuse
* Lower urinary tract obstruction
* Clinically significant anemia or renal dysfunction
* Cardiovascular disease
* Hyperparathyroidism or uncontrolled diabetes
* Generalized skin irritation or significant skin disease
* Use of any medications that could be considered anabolic (e.g. dehydroepiandrosterone (DHEA)) or could interfere with androgen metabolism (e.g. spironolactone, 5-alfa-reductase-inhibitors, ketoconazole, abiraterone)
* Use of estrogens, GnRH agonists/antagonist, antiandrogens, human GH (within previous 12 months of screening)
* Use of testosterone products (within 8 weeks of screening for parenteral products, or 6 weeks of screening for other preparations)
* Sleep apnea
* Untreated depression
* Subject with a partner who is pregnant or will not use contraception

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- AccuMed Research Associates, Garden City, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one study site in the US. Out of 78 subjects screened, 20 subjects were enrolled in the study.
Pre-assignment Details: Apart from having history of hypogonadism, the study subjects were required to present with one or more symptoms of testosterone deficiency (i.e. fatigue, decreased muscle mass, reduced libido, reduced sexual functioning of a non-mechanical nature). The study subjects needed to be in good health despite exhibiting hypogonadism.
Groups:
- Testosterone Topical: Initially subjects self-applied 2.50 mL (two strokes) of testosterone gel by hand every day for seven days followed by a 7-day washout period. After washout period, subjects sequentially self-applied ascending doses of testosterone gel with the applicator; 1.25 mL (one stroke), 2.50 mL (two strokes), and 3.75 mL (three strokes), respectively every day for seven days with no washout period in between.
Period: Overall Study
Arm/Group | Testosterone Topical
Started | 20
Hand Application (2.50 mL) | 20
Washout Period | 20
Applicator Application (1.25 mL) | 19 (One subject discontinued due to non-compliance.)
Applicator Application (2.50 mL) | 18 (One subject discontinued due to physician's decision.)
Applicator Application (3.75 mL) | 18
Completed | 18
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Population: The data are presented for Intent-to-treat (ITT) population, which comprised of all subjects who received at least one dose of the Investigational Medicinal Product (IMP).
Groups:
- Testosterone Topical: Initially study subjects self-applied 2.50 mL (two strokes) of testosterone gel by hand every day for seven days followed by a 7-day washout period. After washout period, study subjects sequentially self-applied ascending doses of testosterone gel with the applicator; 1.25 mL (one stroke), 2.50 mL (two strokes), and 3.75 mL (three strokes), respectively every day for seven days with no washout period in between.
Arm/Group | Testosterone Topical
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Year] | 52.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: subjects]
  United States | 20
Height [Mean (Standard Deviation); unit: inch] | 69.2 (2.7)
Weight [Mean (Standard Deviation); unit: lbs] | 203.7 (29.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate: Percentage of Subjects Whose Average Steady State Concentration (Cavg) of Serum Total Testosterone Levels Are Between 300 and 1050 ng/dL Following Treatment With Each of Three Volumes of FE 999303 Applied With an Applicator.
Description: Descriptive statistics was used to present the outcome results.
Time Frame: Days 15-21, Days 22-28 & Days 29-35
Population: Full Analysis Set (FAS) population was used for this analysis, which comprised of all subjects who had any available Pharmacokinetic (PK) data.
Measure: Number; unit: percentage of subjects
Groups:
- Testosterone 1.25 mL (Applicator): Subjects in this arm self-applied one stroke (1.25 mL) of testosterone gel by applicator to the shoulder/upper arm everyday for seven days.
- Testosterone 2.50 mL (Applicator): Subjects in this arm self-applied two strokes (2.50 mL) of testosterone gel by applicator, one stroke to the shoulder/upper arm and a second stroke to the contralateral shoulder/upper arm everyday for seven days.
- Testosterone 3.75 mL (Applicator): Subjects in this arm self-applied three strokes (3.75 mL) of testosterone gel by applicator, one stroke to the shoulder/upper arm and a second stroke to the contralateral shoulder/upper arm and a third stroke to the first shoulder/upper arm, everyday for seven days.
Arm/Group | Testosterone 1.25 mL (Applicator) | Testosterone 2.50 mL (Applicator) | Testosterone 3.75 mL (Applicator)
Number analyzed (Participants) | 18 | 18 | 18
percentage of subjects | 16.7 | 50.0 | 77.8

2. Secondary Outcome: Responder Rate: Percentage of Subjects Whose Cavg Serum Total Testosterone Levels Are Between 300 and 1050 ng/dL Following Treatment With One Volume of FE 999303 Applied by Hand.
Time Frame: Days 1-7
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Number; unit: percentage of subjects
Groups:
- Testosterone 2.50 mL (Hand): Subjects in this arm self-applied two strokes (2.50 mL) of testosterone gel by hand, one stroke to the shoulder/upper arm and a second stroke to the contralateral shoulder/upper arm everyday for seven days.
Arm/Group | Testosterone 2.50 mL (Hand)
Number analyzed (Participants) | 20
percentage of subjects | 50

3. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT (Dihydrotestosterone) Measuring Area Under the Concentration-time Curve From the Last Dose and 24 Hrs. Post Dose (AUCτ)
Time Frame: Samples were collected pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Day 21, Day 28 & Day 35 of testosterone gel application through applicator
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Mean (Standard Deviation); unit: ng*hr/dL
Arm/Group | Testosterone 1.25 mL (Applicator) | Testosterone 2.50 mL (Applicator) | Testosterone 3.75 mL (Applicator)
Number analyzed (Participants) | 19 | 18 | 18
ng*hr/dL
  Testosterone | 5768 (1228) | 7686 (2648) | 10295 (3764)
  DHT | 688 (349) | 974 (674) | 1223 (666)

4. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Time of Maximum Observed Concentration (Tmax)
Time Frame: as for outcome 3
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Median (Full Range); unit: hr
Arm/Group | Testosterone 1.25 mL (Applicator) | Testosterone 2.50 mL (Applicator) | Testosterone 3.75 mL (Applicator)
Number analyzed (Participants) | 19 | 18 | 18
hr
  Testosterone | 3.77 [0.0 to 24.0] | 3.77 [1.75 to 7.77] | 3.77 [1.77 to 9.92]
  DHT | 3.75 [0.0 to 24.0] | 3.78 [0.0 to 7.77] | 3.86 [1.78 to 24.0]

5. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Maximum Concentration Observed (Cmax)
Time Frame: as for outcome 3
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone 1.25 mL (Applicator) | Testosterone 2.50 mL (Applicator) | Testosterone 3.75 mL (Applicator)
Number analyzed (Participants) | 19 | 18 | 18
ng/dL
  Testosterone | 396 (137) | 641 (319) | 1024 (700)
  DHT | 37.6 (20.3) | 57.7 (39.0) | 78.9 (58.3)

6. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Cavg
Time Frame: as for outcome 3
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone 1.25 mL (Applicator) | Testosterone 2.50 mL (Applicator) | Testosterone 3.75 mL (Applicator)
Number analyzed (Participants) | 19 | 18 | 18
ng/dL
  Testosterone | 240 (51) | 320 (110) | 429 (157)
  DHT | 28.7 (14.5) | 40.6 (28.2) | 51.0 (27.7)

7. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Minimum Concentration Observed (Cmin)
Time Frame: as for outcome 3
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone 1.25 mL (Applicator) | Testosterone 2.50 mL (Applicator) | Testosterone 3.75 mL (Applicator)
Number analyzed (Participants) | 19 | 18 | 18
ng/dL
  Testosterone | 173 (47) | 213 (69) | 250 (116)
  DHT | 21.1 (9.0) | 29.9 (21.9) | 37.3 (22.9)

8. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Time of Minimum Observed Concentration (Tmin)
Time Frame: as for outcome 3
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Median (Full Range); unit: hr
Arm/Group | Testosterone 1.25 mL (Applicator) | Testosterone 2.50 mL (Applicator) | Testosterone 3.75 mL (Applicator)
Number analyzed (Participants) | 19 | 18 | 18
hr
  Testosterone | 7.78 [0.0 to 24.0] | 10.81 [0.0 to 24.0] | 4.76 [0.0 to 24.0]
  DHT | 9.83 [0.0 to 11.8] | 11.0 [0.0 to 24.0] | 9.79 [0.0 to 24.0]

9. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring AUCτ
Time Frame: Samples were collected pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Day 7 of testosterone gel application through hand
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Mean (Standard Deviation); unit: ng*hr/dL
Arm/Group | Testosterone 2.50 mL (Hand)
Number analyzed (Participants) | 20
ng*hr/dL
  Testosterone | 7809 (2609)
  DHT | 1143 (740)

10. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Tmax
Time Frame: as for outcome 9
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Median (Full Range); unit: hr
Arm/Group | Testosterone 2.50 mL (Hand)
Number analyzed (Participants) | 20
hr
  Testosterone | 1.86 [0.0 to 11.8]
  DHT | 1.86 [0.0 to 7.77]

11. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Cmax
Time Frame: as for outcome 9
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone 2.50 mL (Hand)
Number analyzed (Participants) | 20
ng/dL
  Testosterone | 517 (381)
  DHT | 69.1 (58.1)

12. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Cavg
Time Frame: as for outcome 9
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone 2.50 mL (Hand)
Number analyzed (Participants) | 20
ng/dL
  Testosterone | 325 (109)
  DHT | 47.6 (30.8)

13. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Cmin
Time Frame: as for outcome 9
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone 2.50 mL (Hand)
Number analyzed (Participants) | 20
ng/dL
  Testosterone | 234 (62)
  DHT | 35.4 (19.0)

14. Secondary Outcome: Pharmacokinetics of Total Testosterone and DHT Measuring Tmin
Time Frame: as for outcome 9
Population: FAS population was used for this analysis, which comprised of all subjects who had any available PK data.
Measure: Median (Full Range); unit: hr
Arm/Group | Testosterone 2.50 mL (Hand)
Number analyzed (Participants) | 20
hr
  Testosterone | 8.84 [0.0 to 24.0]
  DHT | 11.8 [0.0 to 24.0]

ADVERSE EVENTS:
Time Frame: Overall Treatment Period (36 Days)
Description: Adverse events with onset after start of the first IMP administration were considered treatment-emergent and are presented.
Arm/Group | Testosterone 2.50 mL (Hand) | Testosterone 1.25 mL (Applicator) | Testosterone 2.50 mL (Applicator) | Testosterone 3.75 mL (Applicator)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone 2.50 mL (Hand) (N=20) | Testosterone 1.25 mL (Applicator) (N=20) | Testosterone 2.50 mL (Applicator) (N=20) | Testosterone 3.75 mL (Applicator) (N=20)
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is a restriction on joint publications prepared in collaboration between investigator and sponsor as Ferring reserves the right to be involved in this decision. In the event of any disagreement in the content of any publication both investigator's and Ferring´s opinion will be fairly and sufficiently represented in the publication.